CLINICAL TRIAL: NCT07300839
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED CLINICAL STUDY EVALUATING THE SAFETY, TOLERABILITY, IMMUNOGENICITY AND EFFICACY OF A VARIANT-ADAPTED BNT162B2 VACCINE IN HEALTHY PARTICIPANTS 50 THROUGH 64 YEARS OF AGE
Brief Title: A Study to Learn About a COVID-19 Vaccine in Healthy Adults 50 Through 64 Years of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4591081
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: COVID-19; SARS-COV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BNT162b2 Vaccine (Experimental)
  Interventions: Biological: BNT162b2 Vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BNT162b2 Vaccine — Single dose
  Arms: BNT162b2 Vaccine
Biological: Placebo — Single dose
  Arms: Placebo

SUMMARY:
This study is designed to find out how well the COVID-19 vaccine protects people 50 to 64, who don't have any serious health problems, compared to a group that receives a vaccine that doesn't contain an ingredient to protect against COVID-19 (placebo).

DETAILED DESCRIPTION:
The study is designed to evaluate if the COVID-19 vaccine reduces COVID-19 disease as compared to placebo given to healthy adults 50 to 64 years of age. Approximately 25,500 participants will be randomly chosen to get either one dose of COVID-19 vaccine or of a placebo.

ELIGIBILITY:
Key Inclusion Criteria

* People who are between 50 and 64 years old at their first appointment.
* People who are healthy and, based on their medical history and a doctor's judgment, are considered suitable to join the study.

Key Exclusion Criteria

* People who had COVID-19 in the past 3 months (90 days) before their first visit.
* People who got a COVID-19 vaccine, either as part of a research study or an approved vaccine, in the last 3 months-or plans to get one during the study.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25500 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting local reactions or systemic events | From Day 1 up to 7 days after Vaccination
Percentage of participants reporting adverse events | From Day 1 through 4 weeks after vaccination
Percentage of participants reporting serious adverse events | From Day 1 through 6 months after vaccination
First episode of confirmed COVID-19 cases | From 0 days after vaccination through end of COVID-19 surveillance at least 6 months post-vaccination

SECONDARY OUTCOMES:
First episode of confirmed COVID-19 cases | From 7 days after vaccination through end of COVID-19 surveillance at least 6 months post-vaccination
Geometric Mean Ratio (GMR) | From before vaccination to 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (206):
- United States (206):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - North Alabama Research Center, Athens, Alabama
  - Simon Williamson Clinic / Synexus Clinical Research US, Inc., Birmingham, Alabama
  - Accel Research Sites - Birmingham Clinical Research Unit, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - AMR Clinical, Daphne, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - AMR Clinical, Mobile, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Synexus Clinical Research US, Inc., Phoenix, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Epic Medical Research-Sun City, Sun City, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Synexus Clinical Research US, Inc./Orange Grove Family Practice, Tucson, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Velocity Clinical Research, Chula Vista, Chula Vista, California
  - West Coast Research, Dublin, California
  - Leading Edge Research LA, Encino, California
  - Leading Edge Research, Encino, California
  - Triallogix Medical Corporation, Fullerton, California
  - Marvel Clinical Research, Huntington Beach, California
  - Eximia Research-CA, LLC, La Mesa, California
  - Velocity Clinical Research, Los Angeles, Los Angeles, California
  - ImmuniMet, Modesto, California
  - Carbon Health - North Hollywood - NoHo West, North Hollywood, California
  - Empire Clinical Research, Pomona, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Northern California Research - Sacramento, Sacramento, California
  - Velocity Clinical Research, San Bernardino, San Bernardino, California
  - Artemis Institute for Clinical Research, San Diego, California
  - UCSD AntiViral Research Center (AVRC), San Diego, California
  - Med Partners, Inc. dba Premiere Medical Center of Burbank, Inc., Toluca Lake, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Legacy Clinical Trials, Colorado Springs, Colorado
  - Tekton Research, LLC., Fort Collins, Colorado
  - Tekton Research, LLC., Longmont, Colorado
  - Paradigm Clinical Research, LLC, Wheat Ridge, Colorado
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Clinical Research Consulting, Milford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Washington Health Institute, Washington D.C., District of Columbia
  - Tampa Bay Medical Research, Clearwater, Florida
  - Pioneer Clinical Studies - Coral Gables, Coral Gables, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - Universal Axon Clinical Research, LLC, Doral, Florida
  - Suncoast Research Associates, Doral, Florida
  - AMR Clinical, Fort Myers, Florida
  - Robert B. Pritt, DO, Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Las Mercedes Medical Research, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness, Jupiter, Florida
  - M3 Wake Research - Lake City, Lake City, Florida
  - Accel Research Sites - Lakeland Clinical Research Unit, Lakeland, Florida
  - SRA Trials North, Lauderdale Lakes, Florida
  - Accel Research Sites - Maitland Clinical Research Unit, Maitland, Florida
  - South Florida Research Organization, Medley, Florida
  - Optimal Research, Melbourne, Florida
  - Flourish Research - Miami, LLC, Miami, Florida
  - Florida Pharmaceutical Research & Associates, Inc., Miami, Florida
  - Florida Pharmaceutical Research and Associates, Miami, Florida
  - Nuren Medical and Research Center, Miami, Florida
  - Advanced Clinical Research - Miami - Southwest 92nd Street, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - IMIC, Inc., Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - 3Sync - Hialeah, Miami Lakes, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Angels Clinical Research Institute, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Clinical Neuroscience Solutions - Orlando - South Delaney Avenue, Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - 3SYNC Research - Palm Springs, Palm Springs, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Tropical Clinical Trials, Palmetto Bay, Florida
  - Suncoast Research Associates, Pembroke Pines, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - International Clinical Research - Sanford, Sanford, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Angels Clinical Research Institute, Tampa, Florida
  - Santos Research Center, Tampa, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - DelRicht Research, Atlanta, Georgia
  - AGILE Clinical Research Trials, LLC, Sandy Springs, Georgia
  - M3 Wake Research - Atlanta, Sandy Springs, Georgia
  - Javara - Privia Medical Group Georgia - Savannah, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Chicago Clinical Research Institute, Chicago, Illinois
  - DM Clinical Research - Chicago, Melrose Park, Illinois
  - Koch Family Medicine, Morton, Illinois
  - Accellacare - DuPage, Oak Lawn, Illinois
  - The South Bend Clinic, LLC, South Bend, Indiana
  - University of Iowa, Iowa City, Iowa
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - AMR Clinical, El Dorado, Kansas
  - Johnson County Clinical Trials, Lenexa, Kansas
  - AMR Clinical, Newton, Kansas
  - AMR Clinical, Wichita, Kansas
  - Tekton Research, LLC., Wichita, Kansas
  - AMR Clinical, Lexington, Kentucky
  - DelRicht Research, New Orleans, Louisiana
  - Velocity Clinical Research - New Orleans, New Orleans, Louisiana
  - Pharmaron, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - DM Clinical Research - Boston, Brookline, Massachusetts
  - Walgreens Clinical Trials - Malden, MA, Malden, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Henry Ford St. John Hospital, Grosse Pointe Woods, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - Revival Research Institute, LLC, Southfield, Michigan
  - DM Clinical Research - Detroit, Southfield, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Velocity Clinical Research, Gulfport, Gulfport, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Be Well Clinical Studies - Lincoln, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - McGill Family Practice, Papillion, Nebraska
  - M3 Wake Research - Las Vegas Wellness Way, Las Vegas, Nevada
  - DM Clinical Research - Jersey City, Jersey City, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - DM Clinical Research - Albuquerque, Albuquerque, New Mexico
  - Axces Research, Santa Fe, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Accellacare - Cary, Cary, North Carolina
  - Javara - Tryon Medical Partners, Charlotte, North Carolina
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Accellacare - Hickory, Hickory, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lucas Research, Inc., New Bern, North Carolina
  - Eximia Research - NC, LLC, Raleigh, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Accellacare - Rocky Mount, Rocky Mount, North Carolina
  - Accellacare - Salisbury, Salisbury, North Carolina
  - Accellacare - Piedmont, Statesville, North Carolina
  - Trial Management Associates - Wilmington - Floral Parkway, Wilmington, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Epic Medical Research - Oklahoma, Chickasha, Oklahoma
  - Tekton Research, LLC., Edmond, Oklahoma
  - Tekton Research, LLC., Moore, Oklahoma
  - AMR Clinical, Norman, Oklahoma
  - Tekton Research, LLC., Yukon, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Central Erie Primary Care, Erie, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Trial Management Associates, LLC, Myrtle Beach, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - M3 Wake Research - Chattanooga, Chattanooga, Tennessee
  - AMR Clinical, Knoxville, Tennessee
  - Accellacare US Inc., d/b/a Accellacare of Knoxville, Knoxville, Tennessee
  - Elligo Clinical Research Center, Austin, Texas
  - Orion Clinical Research, Austin, Texas
  - Velocity Clinical Research, Austin, Austin, Texas
  - Headlands Horizons, LLC dba Headlands Research-Brownsville, Brownsville, Texas
  - Epic Medical Research - Carrollton, Carrollton, Texas
  - Lonestar Clinical Research - Dallas, Dallas, Texas
  - Headlands Research-El Paso, El Paso, Texas
  - Cedar Health Research - Euless, Euless, Texas
  - Mercury Clinical Research (Administrative Office), Houston, Texas
  - DM Clinical Research- Cyfair, Houston, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - Mercury Clinical Research - Santa Clara Family Clinic, Houston, Texas
  - DM Clinical Research - Dallas, Irving, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Epic Medical Research - Mesquite, Mesquite, Texas
  - LinQ Research, Pearland, Texas
  - ACRC Trials, Plano, Texas
  - Delricht Research - Prosper: Gen Med, Prosper, Texas
  - Benchmark Research, San Angelo, Texas
  - DM Clinical Research - San Antonio, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - DM Clinical Research - Sugar Land, Sugar Land, Texas
  - Sugar Lakes Family Practice, PA, Sugar Land, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - Cope Family Medicine / CCT Research, Bountiful, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - South Ogden Family Medicine/ CCT Research, South Ogden, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - AMR Clinical, Norfolk, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Tidewater Clinical Research, Virginia Beach, Virginia
  - Eastside Research Associates, Redmond, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591081